CLINICAL TRIAL: NCT01972152
Title: A RANDOMIZED, PHASE 2, DOUBLE-BLIND, 3-WAY CROSSOVER STUDY WITH G-PEN™ (GLUCAGON INJECTION) TO EVALUATE SAFETY, TOLERABILITY AND COMPARATIVE PHARMACOKINETICS AND PHARMACODYNAMICS TO LILLY GLUCAGON™ (GLUCAGON FOR INJECTION [rDNA ORIGIN]) IN HEALTHY VOLUNTEERS
Brief Title: Safety, Tolerability, Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of G-Pen(TM) (Glucagon Injection) to Treat Severe Hypoglycemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Emissary International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XSGP-201; 2R44DK085809-02 (NIH)
Record Dates: First submitted 2013-10-18; First posted 2013-10-30 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Glucagon
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- G-Pen(TM) 1 mg (Experimental): G-Pen(TM) (glucagon injection), single 1 mg subcutaneous (SC) injection
  Interventions: Drug: G-Pen(TM) 1 mg; Drug: Lilly Glucagon(TM) 1 mg; Drug: G-Pen(TM) 0.5 mg
- G-Pen(TM) 0.5 mg (Experimental): G-Pen(TM) (glucagon injection), single 0.5 mg SC injection
  Interventions: Drug: G-Pen(TM) 1 mg; Drug: Lilly Glucagon(TM) 1 mg; Drug: G-Pen(TM) 0.5 mg
- Lilly Glucagon(TM) 1 mg (Active Comparator): Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection
  Interventions: Drug: G-Pen(TM) 1 mg; Drug: Lilly Glucagon(TM) 1 mg; Drug: G-Pen(TM) 0.5 mg

INTERVENTIONS:
Drug: G-Pen(TM) 1 mg
Drug: Lilly Glucagon(TM) 1 mg
Drug: G-Pen(TM) 0.5 mg

SUMMARY:
The purpose of this study is to demonstrate that G-Pen(TM) glucagon is comparable to Lilly Glucagon(TM) in terms of safety and efficacy, as a treatment for severe hypoglycemia, a complication of diabetes.

DETAILED DESCRIPTION:
Primary objective: To Evaluate the Safety and Tolerability of G-Pen™ (Glucagon Injection) 1 mg

Secondary objective (1): To Evaluate the pharmacodynamics (Efficacy) of G-Pen™ (Glucagon Injection) 1 mg

Secondary objective (2):To compare the pharmacokinetics of G-Pen™ (glucagon injection) 1mg [test] administered as 0.5 mg and 1 mg injections, versus Lilly Glucagon™ (glucagon for injection [rDNA origin]) 1 mg (reference)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between the ages of 18 and 60 years of age, inclusive, at Screening.
2. Women must be of non-childbearing potential as defined by one of the following:

   * Females who are >45 and < 60 years of age at Screening and amenorrheic for at least 2 years
   * Females who have had a documented hysterectomy and/or bilateral oophorectomy.
3. Females of childbearing potential with a negative pregnancy test at Screening and Treatment visits, using one of the following forms of contraception for the duration of participation in the study (i.e., until Follow-up 7-14 days post last dose):

   * Oral contraceptive
   * Injectable progesterone
   * Subdermal implant
   * Spermicidal foam/gel/film/cream/suppository
   * Diaphragm with spermicide
   * Copper or hormonal containing intrauterine device (IUD)
   * Sterile male partner vasectomized > 6 month pre-dosing.
4. Male subjects are required to use a condom and one of the methods of contraception in 2. or 3. above starting at Randomization and for the duration of the study.
5. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
6. Subjects must be willing and able to comply with scheduled visits, treatment, laboratory tests and study procedures.

Exclusion Criteria:

1. Recent (i.e., within three (3) months prior to Screening) evidence or medical history of unstable concurrent disease such as: documented evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, immunological, or clinically significant neurological disease.
2. Mean of triplicate set of seated BP readings at Screening, confirmed by 1 set of triplicate at Screening, if deemed necessary where systolic blood pressure (SBP) <90 or >140 mm Hg, and diastolic blood pressure (DBP) <50 or >90 mm Hg.
3. Cardiovascular event within 6 months prior to screening such as unstable angina, acute coronary syndrome, myocardial infarction, therapeutic coronary procedure (e.g., stent placement, Percutaneous Transluminal Coronary Angioplasty (PTCA), Coronary Artery By-pass Grafting (CABG)), stroke or transient ischemic attack.
4. Clinically significant ECG abnormalities.
5. Study participants who are pregnant at Screening are not eligible for this study.
6. Breast feeding must be discontinued if a subject wishes to participate in this study.
7. Positive test for hepatitis B, hepatitis C, or HIV found at Screening.
8. Positive urine drug test for illicit drugs at Screening.
9. Allergies to glucagon, glucagon-like products or to any of the excipients in the investigational formulation.
10. Recent (i.e., within three (3) months prior to Screening) administration of glucagon.
11. Any prior cerebrovascular accident or major permanent neurological damage such as aphasia, hemiparesis, or dementia.
12. Peripheral artery disease with uncontrolled claudication
13. Current diagnosis or current clinical evidence of any New York Heart Association classification of heart failure.
14. Subjects with any of the following abnormalities in clinical laboratory tests at Screening, confirmed by a single repeat, if necessary:

    * Total bilirubin > 1.5x upper limit of normal (ULN)
    * aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) ≥ 2.5x ULN.
    * Creatinine > 2.5x ULN.
15. History of regular alcohol consumption as defined by alcohol intake in a quantity exceeding 7 drinks per week for females or 14 drinks per week for males, where 1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor.
16. Participation in other studies involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before screening for the current study and during participation in the current study.
17. Blood donation of approximately 1 pint (500 mL) within 8 weeks prior to Screening.
18. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — Texas Diabetes Institute, University Health System
Locations (1):
- Texas Diabetes Institute, University Health System, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study involved healthy volunteers who were recruited from the local community surrounding a state-affiliated diabetes treatment center over a period of 3 months.
Pre-assignment Details: Of a total of 41 individuals recruited, 4 declined participation, 7 did not meet eligibility criteria and 30 were enrolled.
Groups:
- G-Pen(TM) 0.5 mg First, Then G-Pen(TM) 1 mg, Then Lilly 1 mg: G-Pen(TM) (glucagon injection), single 0.5 mg subcutaneous (SC) injection at treatment visit 1 followed by a 3-14 day washout, G-Pen(TM) (glucagon injection), single 1 mg subcutaneous (SC) injection at treatment visit 2 followed by a 3-14 day washout, Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection at treatment visit 3.
- G-Pen(TM) 0.5 mg First, Then Lilly 1 mg, Then G-Pen(TM) 1 mg: G-Pen(TM) (glucagon injection), single 0.5 mg subcutaneous (SC) injection at treatment visit 1 followed by a 3-14 day washout, Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection at treatment visit 2, G-Pen(TM) (glucagon injection), single 1 mg subcutaneous (SC) injection at treatment visit 3.
- G-Pen(TM) 1 mg First, Then G-Pen(TM) 0.5 mg , Then Lilly 1 mg: G-Pen(TM) (glucagon injection), single 1 mg subcutaneous (SC) injection at treatment visit 1 followed by a 3-14 day washout, G-Pen(TM) (glucagon injection), single 0.5 mg SC injection at treatment visit 2 followed by a 3-14 day washout, Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection at treatment visit 3.
- G-Pen(TM) 1 mg First, Then Lilly 1 mg, Then G-Pen(TM) 0.5 mg: G-Pen(TM) (glucagon injection), single 1 mg subcutaneous (SC) injection at treatment visit 1 followed by a 3-14 day washout, Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection of at treatment visit 2 followed by a 3-14 day washout, G-Pen(TM) (glucagon injection), single 0.5 mg SC injection at treatment visit 3.
- Lilly 1 mg First, Then G-Pen(TM) 0.5 mg, Then G-Pen(TM) 1 mg: Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection at treatment visit 1 followed by a 3-14 day washout, G-Pen(TM) (glucagon injection), single 0.5 mg subcutaneous (SC) injection at treatment visit 2 followed by a 3-14 day washout, G-Pen(TM) (glucagon injection), single 1 mg subcutaneous (SC) injection at treatment visit 3.
- Lilly 1 mg First, Then G-Pen(TM) 1 mg, Then G-Pen(TM) 0.5 mg: Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection at treatment visit 1 followed by a 3-14 day washout, G-Pen(TM) (glucagon injection), single 1 mg subcutaneous (SC) injection at treatment visit 2 followed by a 3-14 day washout, G-Pen(TM) (glucagon injection), single 0.5 mg subcutaneous (SC) injection at treatment visit 3.
Period: First Treatment Visit
Arm/Group | G-Pen(TM) 0.5 mg First, Then G-Pen(TM) 1 mg, Then Lilly 1 mg | G-Pen(TM) 0.5 mg First, Then Lilly 1 mg, Then G-Pen(TM) 1 mg | G-Pen(TM) 1 mg First, Then G-Pen(TM) 0.5 mg , Then Lilly 1 mg | G-Pen(TM) 1 mg First, Then Lilly 1 mg, Then G-Pen(TM) 0.5 mg | Lilly 1 mg First, Then G-Pen(TM) 0.5 mg, Then G-Pen(TM) 1 mg | Lilly 1 mg First, Then G-Pen(TM) 1 mg, Then G-Pen(TM) 0.5 mg
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 4 | 5 | 5 | 5 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Period: Second Treatment Visit
Arm/Group | G-Pen(TM) 0.5 mg First, Then G-Pen(TM) 1 mg, Then Lilly 1 mg | G-Pen(TM) 0.5 mg First, Then Lilly 1 mg, Then G-Pen(TM) 1 mg | G-Pen(TM) 1 mg First, Then G-Pen(TM) 0.5 mg , Then Lilly 1 mg | G-Pen(TM) 1 mg First, Then Lilly 1 mg, Then G-Pen(TM) 0.5 mg | Lilly 1 mg First, Then G-Pen(TM) 0.5 mg, Then G-Pen(TM) 1 mg | Lilly 1 mg First, Then G-Pen(TM) 1 mg, Then G-Pen(TM) 0.5 mg
Started | 5 | 4 | 5 | 5 | 5 | 5
Completed | 5 | 3 | 5 | 5 | 5 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Period: Third Treatment Visit
Arm/Group | G-Pen(TM) 0.5 mg First, Then G-Pen(TM) 1 mg, Then Lilly 1 mg | G-Pen(TM) 0.5 mg First, Then Lilly 1 mg, Then G-Pen(TM) 1 mg | G-Pen(TM) 1 mg First, Then G-Pen(TM) 0.5 mg , Then Lilly 1 mg | G-Pen(TM) 1 mg First, Then Lilly 1 mg, Then G-Pen(TM) 0.5 mg | Lilly 1 mg First, Then G-Pen(TM) 0.5 mg, Then G-Pen(TM) 1 mg | Lilly 1 mg First, Then G-Pen(TM) 1 mg, Then G-Pen(TM) 0.5 mg
Started | 5 | 3 | 5 | 5 | 5 | 5
Completed | 5 | 3 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study involved a 3-way cross-over design with 30 total randomized subjects, so the baseline characteristics are the same for all 3 arms.
Groups:
- Total Study Group: Includes all 30 randomized subjects
Arm/Group | Total Study Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Number of serious adverse events (SAEs) per treatment group
Time Frame: From first dose until completion of the post-treatment follow-up visit, up to 6 weeks
Population: All subjects receiving treatment were included in this analysis.
Measure: Number; unit: events
Groups:
- G-Pen(TM) 1 mg: G-Pen(TM) (glucagon injection), single 1 mg SC injection
  G-Pen(TM) 1 mg
  Lilly Glucagon(TM) 1 mg
  G-Pen(TM) 0.5 mg
- G-Pen(TM) 0.5 mg: G-Pen(TM) (glucagon injection), single 0.5 mg SC injection
  G-Pen(TM) 1 mg
  Lilly Glucagon(TM) 1 mg
  G-Pen(TM) 0.5 mg
- Lilly Glucagon(TM) 1 mg: Lilly Glucagon(TM) [glucagon for injection (rDNA origin)], single 1 mg SC injection
  G-Pen(TM) 1 mg
  Lilly Glucagon(TM) 1 mg
  G-Pen(TM) 0.5 mg
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 29 | 28
events | 0 | 0 | 0

2. Secondary Outcome: Glucose Area Under the Curve (AUC)
Description: Pharmacodynamic parameter: Glucose area under the curve from baseline to 240 minutes post-treatment
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: Per protocol analysis set. Two subjects were excluded from all analyses: one who completed no treatment visits and had no evaluable data and another who violated eligibility criteria. A third subject was excluded from analysis for the one treatment visit at which the subject's blood samples were inadvertently diluted with saline during collection.
Measure: Mean (Standard Deviation); unit: min*mg/dL
Groups:
- G-Pen(TM) 1 mg: G-Pen(TM) (glucagon injection), single 1 mg SC injection
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
min*mg/dL | 481.1 (64.9) | 467 (47.9) | 473.5 (72.9)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.24, Mixed Models Analysis; Data were log transformed for analysis

3. Secondary Outcome: Glucose Cmax
Description: Pharmacodynamic parameter: Maximum concentration of glucose
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
mg/dL | 148.04 (24.94) | 140.32 (23.59) | 154.9 (28.02)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.34, Mixed Models Analysis — Data were log transformed for analysis
Statistical Analysis 2: Comparison: G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — Data were log transformed for analysis

4. Secondary Outcome: Glucose Tmax
Description: Pharmacodynamic parameter: Time to Maximum Glucose Concentration
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
minutes | 48.2 (11.8) | 44.5 (11.2) | 46.5 (20.5)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.95, Mixed Models Analysis

5. Secondary Outcome: Glucose AUCex
Description: Pharmacodynamic parameter: Area Under the Glucose Excursion Curve
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*mg/dL
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
min*mg/dL | 228.5 (89.1) | 197.3 (74.7) | 223 (101.5)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.76, Mixed Models Analysis

6. Secondary Outcome: Glucose MAE
Description: Pharmacodynamic parameter: Maximum absolute glucose excursion from baseline
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
mg/dL | 50.8 (22) | 42.5 (19.8) | 53.2 (18.8)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.68, Mixed Models Analysis
Statistical Analysis 2: Comparison: G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

7. Secondary Outcome: Glucose Tex
Description: Pharmacodynamic parameter: Earliest reported time of MAE, based on within-subject changes from baseline
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
minutes | 48.2 (11.8) | 61.6 (52.3) | 68.8 (44.4)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis; Data were log transformed for analysis

8. Secondary Outcome: Glucagon AUC
Description: Pharmacokinetic parameter: Glucagon area under the curve from baseline to 240 minutes post-treatment
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*pg/ml
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
min*pg/ml | 3259.9 (3447.5) | 2105.3 (2381.9) | 4781.7 (2222.9)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Data were log transformed for analysis
Statistical Analysis 2: Comparison: G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Data were log transformed for analysis

9. Secondary Outcome: Glucagon Cmax
Description: Pharmacokinetic parameter: Maximum concentration of glucagon
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
pg/ml | 2055.4 (2052) | 1318.8 (1435.8) | 4429.9 (3970)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Data were log transformed for analysis
Statistical Analysis 2: Comparison: G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Data were log transformed for analysis

10. Secondary Outcome: Glucagon Tmax
Description: Pharmacokinetic parameter: Time to maximum concentration of glucagon
Time Frame: Approximately 15 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 240 minutes post-injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Number analyzed (Participants) | 28 | 28 | 27
minutes | 37.6 (15.2) | 33.3 (13.2) | 18.9 (10.1)
Statistical Analysis 1: Comparison: G-Pen(TM) 1 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: G-Pen(TM) 0.5 mg vs Lilly Glucagon(TM) 1 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first administration of study drug to an untreated follow-up visit occurring 7-14 days after the last treatment, up to 6 weeks.
Description: Adverse events are reported by Preferred Term
Arm/Group | G-Pen(TM) 1 mg | G-Pen(TM) 0.5 mg | Lilly Glucagon(TM) 1 mg
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 22/28 | 26/29 | 22/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Pen(TM) 1 mg (N=28) | G-Pen(TM) 0.5 mg (N=29) | Lilly Glucagon(TM) 1 mg (N=28)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (5) | 13 (14)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Flushing (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Hot Flushes (Endocrine disorders) | 0 (0) | 1 (1) | 3 (3)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 21 (25) | 24 (32) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No